CLINICAL TRIAL: NCT02866357
Title: Multiplex Molecular Detection of Respiratory Pathogens of Adult Patients Admitted to Hospital for Exacerbation of Asthma and Chronic Obstructive Pulmonary Disease and Their Clinical Outcomes.
Brief Title: Respiratory Pathogens of Patients With Asthma and COPD Exacerbations
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fanny W.S. Ko, Honorary Associate Professor, Chinese University of Hong Kong
Other Study IDs: COPD-asthma microb_v02
Record Dates: First submitted 2016-08-10; First posted 2016-08-15 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasopharyngeal aspirate
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention — Just collection of nasopharyngeal aspirate for assessment

SUMMARY:
To assess the infective etiologies by quantitative polymerase chain reaction (qPCR) of acute exacerbation of COPD and asthma who required hospitalization.

To identify the HRV subtypes that are associated with COPD and asthmaexacerbations.

To assess if the infective aetiologies have associations with the clinical outcome of the patients.

DETAILED DESCRIPTION:
Objective: Chronic obstructive pulmonary disease (COPD) and asthma exacerbations both contribute to significant health care burden. Viral infections are important cause of acute exacerbation of COPD and asthma.

Hypothesis to be tested: 1. Assess infective etiologies by Multiplex Molecular Detection of nasopharyngeal aspirate (NPA) of patients with acute exacerbation of COPD and asthma; 2. Identify the human rhinovirus (HRV) (the commonest virus causing exacerbations) subtypes involved; 3.Assess if the infective etiologies have associations with clinical outcome of the patients.

Design and subjects: Prospective observational study. Patients admitted to hospital for acute exacerbation of COPD and asthma. Stable COPD and asthma patients will be recruited as controls.

Study instruments: Multiplex Molecular Detection of respiratory pathogens from NPA. Clinical data of the patient will be collected and spirometry will be performed.

Interventions: NPA collection from subjects. Main outcome measures: Primary aim is assessment of the prevalence of different viruses in relation to acute exacerbation of asthma and COPD. Secondary aim is to assess if a certain pathogen is associated with clinical outcomes including duration of hospitalization and 30 and 60 day readmissions and mortality Data analysis: Data will be analyzed by the Statistical Package of the Social Science Statistical software for Window, Version 22 (IBM SPSS Inc, IL, USA). Statistical methods including chi-square test, student t test and ANOVA will be used as appropriate.

Expected results: Understanding the epidemiology of respiratory viruses in COPD and asthma exacerbations allows further investigations of treatment options and gives information about the prognosis.

ELIGIBILITY:
Inclusion Criteria:

For COPD patients, patients who are admitted to the Prince of Wales Hospital with AECOPD will be screened for this study. AECOPD is defined when a patient with background COPD (with lung function parameters of FEV1/FVC ratio <70%)24 presented with at least two of the following major symptoms (increased dyspnoea, increased sputum purulence, increased sputum volume) or one major and one minor symptom (nasal discharge/congestion, wheeze, sore throat, cough) for at least two consecutive days.25,26

Inclusion criteria:

1. Patients who has background COPD as mentioned above fulfilling the exacerbation criteria
2. Age ≥40 years

For asthma patients, patients who are admitted to the Prince of Wales Hospital with asthma exacerbation will be screened for this study. Acute exacerbation of asthma is defined when an asthma patient presents with increasing dyspnea, wheeze or cough.

Inclusion criteria:

1. Patients who has background asthma (defined as those with a consistent history and prior documented evidence of variable airflow obstruction, with evidence of an increase in FEV1 greater than 12% or 400 mL following bronchodilator or bronchial hyperresponsiveness on bronchial provocation testing, when stable)6 with any of the above exacerbation criteria for at least 2 consecutive days.
2. Age ≥18 years

Control asthma and COPD subjects will be recruited from the respiratory clinic of the Prince of Wales Hospital. Subjects will be matched for age, sex and lung function of the COPD and asthma subjects. All recruited COPD subjects should have FEV1/FVC ratio of <70%. For asthma patients, they should have a clinical diagnosis of asthma (defined as those with a consistent history and prior documented evidence of variable airflow obstruction, with evidence of an increase in FEV1 greater than 12% or 400 mL following bronchodilator or bronchial hyperresponsiveness on bronchial provocation testing, when stable). These subjects should have no exacerbation of asthma or COPD 6 weeks prior to the assessment.

Exclusion Criteria:

Exclusion criteria for all patients:

1. History of lung resection or other significant pulmonary disease like pulmonary fibrosis.
2. Active infection like pulmonary tuberculosis
3. Unable to complete assessment due to physical and/or cognitive impairment
4. Having short life expectancy like subjects with terminal malignancy or intractable heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asthma and COPD patients
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2016-08; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of different types of viruses | 1 month
  Prevalence of different types of viruses

SECONDARY OUTCOMES:
Clincial outcomes | 60 days
  The secondary aim is to assess if a certain pathogen has association with clinical outcomes including duration of hospitalization and 30 and 60 day readmissions and mortality.

CONTACTS AND LOCATIONS:
Overall Officials: David S Hui, MD, Study Chair — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ko FW, Chan PK, Chan RWY, Chan KP, Ip A, Kwok A, Ngai JC, Ng SS, On CT, Hui DS. Molecular detection of respiratory pathogens and typing of human rhinovirus of adults hospitalized for exacerbation of asthma and chronic obstructive pulmonary disease. Respir Res. 2019 Sep 13;20(1):210. doi: 10.1186/s12931-019-1181-0. PMID 31519188